CLINICAL TRIAL: NCT03276000
Title: Randomized Control Trial Comparing Patient Acceptability and Tolerance to Pain Using Oral Versus Vaginal Misoprostol for Cervical Priming Before Office Hysteroscopy.
Brief Title: Misoprostol for Cervical Priming Before Office Hysteroscopy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12345
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Misoprostol Allergy
Keywords: Misoprostol ,office hysteroscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): 50 patients receive 200 mg oral misoprostol (Misotac; Sigma Pharm) 3h before office hysteroscopy
  Interventions: Procedure: office hysteroscopy
- group B (Active Comparator): 50 patients receive 200 mg misoprostol (Misotac; Sigma Pharm) 3h before office hysteroscopy moistened with saline solution will be inserted in posterior fornix of vagina.
  Interventions: Procedure: office hysteroscopy

INTERVENTIONS:
Procedure: office hysteroscopy — A rigid 30 4-mm hysteroscope (Karl Storz Endoscopy) will be used without anaesthesia or analgesia 3 hours after administration of misoprostol. The uterine cavity will be distended with normal saline solution at a pressure of 100-120 mm Hg. The vaginoscopic ''no touch'' technique was followed; no speculum or tenaculum was used.

SUMMARY:
The objective of the present study is to evaluate the appropriate route of administration of misoprostol, either oral or vaginal, for cervical priming to facilitate the procedure of office hysteroscopy and reduce patient discomfort to minimum

DETAILED DESCRIPTION:
Sample size calculation was done using the comparison of pain sensation represented through VAS between oral and vaginal misoprostol for cervical ripening before office hysteroscopy. As reported in previous publication (Sordia-Herna'ndez et al., 2011), the mean ±SD of VAS in oral misoprostol group was approximately 6.04 ± 1.5, while in vaginal misoprostol group was approximately 2.8 ± 1.2. Accordingly, we calculated that the minimum proper sample size was 23 women in each arm to be able to detect a real difference of 1 unit with 80% power at α = 0.05 level using Student's t test for independent samples. Sample size calculation was done using Stats Direct statistical software version 2.7.2 for MS Windows, StatsDirect Ltd., Cheshire, UK

However, the study population consists of 100 patients in reproductive age that requires diagnostic hysteroscopy for investigation of infertility or AUB.

The patients will be recruited from Office hysteroscopy clinic of the Obstetrics and Gynecology Department, Faculty of Medicine, Cairo University from October 2017 to march 2018.

The Patients will be allocated equally into 2 groups ( each group contain 50 patients)

Groups will be as follows:

1. Group A: 50 patients receive 200 mg oral misoprostol (Misotac; Sigma Pharm) 3h before the procedure.
2. Group B: 50 patients receive 200 mg misoprostol (Misotac; Sigma Pharm) 3h before the procedure moistened with saline solution will be inserted in posterior fornix of vagina.

ELIGIBILITY:
Inclusion criteria:

1. Patients indicated for diagnostic hysteroscopy for infertility or AUB.
2. Reproductive age >19 - 45yrs.
3. Postmenstrual between days 7 and 11 of the cycle ( except in irregular bleeding)

Exclusion criteria:

Contraindicating the use of prostaglandins such as:-

1. Cardiovascular disease
2. Severe bronchial asthma.
3. Hypertension.
4. Renal failure.
5. Known sensitivity to Prostaglandins

Contraindication to office hysteroscopy such as:-

1. Pelvic inflammatory disease.
2. Marked cervical stenosis.
3. Known cervical malignancy.
4. pregnancy
5. profuse uterine bleeding
6. Recent uterine perforation.

Neurological disorders affecting the evaluation of pain.

Previous cervical surgery.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain sensation: | The VAS will be applied immediately after the procedure ended.
  the level of pelvic pain will be rated according to a 10-point visual analogue scale (VAS).
Patient acceptability | The VAS will be applied immediately after the procedure ended.
  according to a 10-point VAS

SECONDARY OUTCOMES:
Bleeding | during the procedure.
  Bleeding during and after the procedure.
Procedure time | it will be reported immediately after the process ended
  Procedure time from introduction of the office hysteroscopy through the external cervical os and the visualization of the uterine cavity.
Ease of cervical entry by hysteroscopy | The VAS will be applied immediately after the procedure ended.
  Ease of cervical entry by hysteroscopy to evaluate the uterine cavity according to a 10-point VAS.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sordia-Hernandez LH, Rosales-Tristan E, Vazquez-Mendez J, Merino M, Iglesias JL, Garza-Leal JG, Morales A. Effectiveness of misoprostol for office hysteroscopy without anesthesia in infertile patients. Fertil Steril. 2011 Feb;95(2):759-61. doi: 10.1016/j.fertnstert.2010.07.1066. Epub 2010 Aug 21. PMID 20728083
- [Background] Bastu E, Celik C, Nehir A, Dogan M, Yuksel B, Ergun B. Cervical priming before diagnostic operative hysteroscopy in infertile women: a randomized, double-blind, controlled comparison of 2 vaginal misoprostol doses. Int Surg. 2013 Apr-Jun;98(2):140-4. doi: 10.9738/INTSURG-D-12-00024.1. PMID 23701149
- [Background] El-Mazny A, Abou-Salem N. A double-blind randomized controlled trial of vaginal misoprostol for cervical priming before outpatient hysteroscopy. Fertil Steril. 2011 Oct;96(4):962-5. doi: 10.1016/j.fertnstert.2011.04.049. Epub 2011 May 14. PMID 21575939